CLINICAL TRIAL: NCT02351050
Title: Sonolysis in Risk Reduction of Symptomatic and Silent Brain Infarctions During Coronary Stenting Due to Ultrasound Activation of Endogenous Fibrinolytic System Using Transcranial Doppler Monitoring
Brief Title: Sonolysis in Risk Reduction of Symptomatic and Silent Brain Infarctions During Coronary Stenting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 13595
Record Dates: First submitted 2014-11-23; First posted 2015-01-30 (Estimated); Last update posted 2018-03-26 (Actual); Status verified 2018-03

CONDITIONS: Coronary Artery Disease
Keywords: sonolysis, brain infarction, coronary angioplasty
MeSH Terms: conditions — Coronary Artery Disease; Brain Infarction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sonolysis (Experimental): continual transcranial Doppler monitoring with maximal intensity during endovascular procedure
  Interventions: Device: Sonolysis
- placebo (Placebo Comparator): sham transcranial Doppler monitoring during endovascular procedure
  Interventions: Other: Sham procedure

INTERVENTIONS:
Device: Sonolysis — continual transcranial Doppler monitoring of middle cerebral artery
  Other Names: sonothrombolysis, sonothrombotripsy
  Arms: Sonolysis
Other: Sham procedure — sham transcranial Doppler monitoring of middle cerebral artery
  Arms: placebo

SUMMARY:
The aim of the project is to demonstrate a fibrinolytic effect of sonothrombolysis (continual transcranial Doppler monitoring) using 2 MHz diagnostic probe on the reduction of risk of brain infarctions due to the activation of endogenous fibrinolytic system during angioplasty and stenting of coronary arteries. 120 patients indicated for coronary angioplasty and stenting will be enrolled into the study in order to demonstrate a twenty-percent risk reduction of number and volume of brain infarctions detected using MRI examination 24 hours after cardiac endovascular treatment in 5% level of significance. Patients will be randomized - subgroup 1 will undergo a 40-240 minute non-diagnostic TCD monitoring during endovascular procedure, subgroup 2 will undergo interventions without TCD monitoring.

Confirmation of our hypothesis that sonothrombolysis is able to activate endogenous fibrinolytic system during coronary angioplasty and stenting with consecutive reduction of the number and volume of brain infarcts, can lead to the increase of the safety these patients. We can presume that up to 50% of patients indicated for endovasular heart treatment can be treated using these methods in the future.

DETAILED DESCRIPTION:
AIM OF THE PROJECT The aim of the project is to demonstrate an effect of continual TCD monitoring using 2 MHz diagnostic probe with maximal diagnostic energy on the reduction of risk of brain microinfarctions due to the activation of endogenous fibrinolytic system and mechanical effect on emboli during coronary stenting.

HYPOTHESIS Sonothrombolysis lead to activation of fibrinolytic system in both healthy volunteers and acute stroke patients. In acute stroke patients, mechanical effect of sonothrombolysis is the second effect leading to acceleration of occluded artery recanalization. We hypothesize that combination of mechanical effect and activation of fibrinolytic system during sonothrombolysis (TCD monitoring) during coronary stenting will lead to recanalization of small arterial occlusions caused by microembolization during intervention. The result will be reduction of volume and the number of brain infarctions.

120 patients indicated for coronary stenting will be enrolled into the study in order to demonstrate a twenty-percent risk reduction of number and volume of brain infarctions detected using MRI examination 24 hours after procedure in 5% level of statistical significance. Patients will be randomized into 2 subgroups. Subgroup 1 will undergo non-diagnostic bilateral TCD monitoring during coronary stenting. Subgroup 2 will undergo coronary stenting without TCD monitoring.

PATIENTS AND METHODS Patients: 120 patients indicated for coronary angioplasty and stenting will be enrolled into the study during a 3-year period. All 120 patients will be randomized for standard coronary angioplasty and stenting and TCD monitored.

Clinical examinations: Physical and neurological examinations including evaluating of neurological impairment of neurological deficit in NIHSS scale, modified Rankin scale and cognitive testing (Mini Mental State Examination, Clock drawing test) will be performed before and 24 - 72 hours after coronary angioplasty and stenting.

Randomization: Randomization using computer generated random allocation will be used.

Sonothrombolysis: In patients randomized into sonothrombolysis subgroup, bilateral MCA segment in depth 55 mm will be monitored for 40 - 240 minutes using a diagnostic 2 MHz probe with maximal diagnostic energy. Non-diagnostic TCD monitoring will be performed without detection of microembolic signals or detection of changes in blood flow. The second (control) subgroup will undergo a standard coronary angioplasty and stenting without sonothrombolysis.

MRI protocol will consists of 4 sequences: 1. Localizer; 2. T2TSE; 3. FLAIR; 4. DWI. Sequences 1-3 will be applied in the same level, they will have the same slice thickness and the same cut number. The slice thickness comprises its own cut thickness (5 mm) + distant factor (30%). Standard number of slices is 19. Standard slice level is considered to be a modified level of skull base due to the minimalization of distant artifacts EPI sequence. T2TSE: TR=4000/TE=99/ETL=9, FOV 230, FOV ph. 75%, matrix 256x256. FLAIR: 8050/112/ETL=21/2 conc., FOV 230, FOV ph. 76,6%, matrix 256x151. EPI-DWI: 4200/139/EPI f.=96/6 av., FOV 230, FOV ph. 100%, phase enc. direction A-P, matrix 128x96 with interpolation, phase partial Fourier 6/8, Bw 1346 Hz/Px, echo spacing 0.83 ms, TA. Sequence called "trace" with three types of MR pictures in every slice: (a) T2*EPI b=0; (b) DWI b=500; (c) DWI b=1000. The fourth type of images automatically created an ADC map (in-line postprocessing). DWI show a middle (average) diffusivity of every point of examined brain tissue when b value is 500 and 1000. This sequence is applied in order to assess hemorrhage (T2*EPI) and monitor sites of reduced diffusion (DWI, b=500 and 1000). New infarctions will be evaluated in the all of brain territories.

Adverse effects: All adverse effects during 1 month after UM will be registered, especially all causes for new admissions to the hospital, worsening of neurological symptoms (>4 points in NIH stroke scale), brain edema, symptomatic and asymptomatic intracranial bleeding detected in control brain MRI.

Study protocol has been approved by the Ethics Committees in accordance with the principles and guidelines of the Declaration of Helsinki, 1975.

ELIGIBILITY:
Inclusion Criteria:

* age 35-90 years
* sufficient temporal bone window for TCD with detectable blood flow in MCA
* independent patient (modified Rankin score 0-2)
* informed consent signed by the patient
* coronary angioplasty and stenting will be performed as an elective procedure

Exclusion Criteria:

* contra-indication for MRI examination (pace-maker, implanted metal material, claustrophobia)
* emergent coronary angioplasty and stenting

Ages: 35 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
New infarction | 24 hours after intervention
  New brain infarction detected using magnetic resonance diffusion weighted images (MRI-DWI)

SECONDARY OUTCOMES:
Cognitive functions changes, measured by ADAS, MMSE, Clock Drawing Test and Verbal Fluency Test | 7 and 30 days after interventions
  Cognitive decline measured by ADAS, MMSE, Clock Drawing Test and Verbal Fluency Test
Large new infarction, infarction ≥0.5 mL detected using magnetic resonance diffusion weighted images (MRI-DWI) | 24 hours after intervention
  New brain infarction ≥0.5 mL detected using magnetic resonance diffusion weighted images (MRI-DWI)
Volume of new brain infarction, detected using magnetic resonance diffusion weighted images (MRI-DWI) | 24 hours after intervention
  Volume of new brain infarctions detected using magnetic resonance diffusion weighted images (MRI-DWI)
30-days morbidity and mortality | 30 days after intervention
  stroke, TIA, myocardial infarctions and death during 30 days after intervention
Symptomatic intracerebral hemorrhage, detected using magnetic resonance (MRI) | 24 hours after intervention
  Intracerebral hemorrhage with worsening of neurological status (≥ 4 points in NIHSS scale) detected using magnetic resonance (MRI)

CONTACTS AND LOCATIONS:
Overall Officials: David Skoloudik, MD, Prof, Study Chair — University Hospital Ostrava
Locations (1):
- University Hospital Nitra, Nitra, Slovakia

IPD SHARING:
Plan to Share IPD: Undecided